CLINICAL TRIAL: NCT04878107
Title: SBRT/LDRT in Combination With Camrelizumab and Apatinib in Metastatic Non-small Cell Lung Cancer Patient Previously Treated With PD-1/L1 Inhibitor and Chemotherapy：a Prospective Exploratory Study
Brief Title: SBRT/LDRT in Combination With Camrelizumab and Apatinib in Metastatic Non-small Cell Lung Cancer Patient Previously Treated With PD-1/L1 Inhibitor and Chemotherapy
Acronym: SABRE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, Director of Department of Radiation and Medical Oncology, Wuhan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021061
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: stereotactic body radiotherapy; Low-Dose Radiation Therapy; Camrelizumab; Apatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT/LDRT + Camrelizumab +Apatinib (Experimental): SBRT（8Gy×3f） LDRT（2Gy×5f） Camrelizumab（200mg，q3w） Apatinib （250mg，qd）
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Radiation: SBRT; Radiation: LDRT
- SBRT + docetaxel (Active Comparator): docetaxel 75mg/m2 SBRT（8Gy×3f）
  Interventions: Drug: Docetaxel injection; Radiation: SBRT

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab (AiRuiKa™), a programmed cell death 1 (PD-1) inhibitor being developed by Jiangsu Hengrui Medicine Co. Ltd
  Other Names: SHR1210
  Arms: SBRT/LDRT + Camrelizumab +Apatinib
Drug: Apatinib — Apatinib [Aitan® (brand name in China)], also known as rivoceranib, is a novel, small molecule, selective vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitor
  Arms: SBRT/LDRT + Camrelizumab +Apatinib
Drug: Docetaxel injection — Docetaxel is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug
  Arms: SBRT + docetaxel
Radiation: SBRT — Stereotactic body radiation therapy (SBRT) is a cancer treatment that delivers extremely precise, very intense doses of radiation to cancer cells while minimizing damage to healthy tissue. SBRT involves the use of sophisticated image guidance that pinpoints the exact three-dimensional location of a tumor so that the radiation can be more precisely delivered to cancer cells.
Radiation: LDRT — low dose radation therapy
  Arms: SBRT/LDRT + Camrelizumab +Apatinib

SUMMARY:
SABRE STUDY will explore effectiveness and safety of the combination therapy of camrelizumab，apatinib and SBRT/LDRT in patients with metastatic non-small Cell Lung Cancer (NSCLC) patient previously treated With PD-1/L1 Inhibitor and Chemotherapy.

DETAILED DESCRIPTION:
SABRE STUDY consists of two stages.

first stage of this trial is a single-arm study that requires enrolling at least 18 patients, all of whom would receive the treatment of SBRT/LDRT in combination with apatinib plus camrelizumab.The trial would proceed into the second stage if 4 or more patients achieve CR/PR. Otherwise, the trial is stopped early due to futility as we fail to reject the null.

In the second stage, at least 70 patients are equally randomized into two arms to receive "SBRT/LDRT in combination with apatinib plus camrelizumab" or "SBRT + docetaxel" . Stratified-area group randomization would be used.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell lung cancer（NSCLC）
* Has previous treatment with PD-1/L1 monoclonal antibody in combination with a platinum-based chemotherapy with outcome of complete remission (CR), partial remission (PR), or stable disease (SD) for ≥ 6 months
* Has at least two disseminated lesions for LDRT and SBRT, respectively
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
* Has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) or ROS Proto-Oncogene 1(ROS1)-directed therapy is not indicated
* Has adequate organ function
* For female subjects of childbearing potential, a serum pregnancy test should be performed within 7 days prior to the administration of the first study intervention (study drug, radiation therapy) and have a negative result. Subjects are required to agree to use highly effective contraception (i.e., a method with a failure rate of less than 1% per year) and continue until at least 180 days after discontinuation of trial treatment

Exclusion Criteria:

* Imaging (CT or MRI) shows evidence of tumour invasion of large blood vessels or poorly demarcated blood vessels or the presence of cavities and necrotic lesions in the lungs
* With active bleeding or perforation or a hereditary or acquired bleeding tendency present, with a daily haemoptysis of ≥2.5mL in the 3 months prior to screening.
* with hypertensive disorders that cannot be reduced to the normal range with antihypertensive medication (systolic blood pressure ≤ 140 mmHg / diastolic blood pressure ≤ 90 mmHg).
* Urine routine suggesting urine protein ≥ (++) and 24-hour urine protein amount ≥ 1.0g.
* presence of thrombotic disease requiring long-term anticoagulation with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day).
* Previous systemic antitumour therapy other than PD-1(L1) monoclonal antibody in combination with platinum-based chemotherapy, or previous treatment with anti-angiogenic agents (including bevacizumab, apatinib, anlotinib, etc.).
* Immune-related adverse events in previous PD-1(L1) therapy leading to treatment discontinuation
* Symptomatic, untreated or actively progressing central nervous system (CNS) metastases are confirmed by CT or MRI assessment during screening and prior to radiographic evaluation.
* Subjects with grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval > 450 ms for males and QTc interval > 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% according to NYHA criteria
* Has known history of Human Immunodeficiency Virus (HIV)
* Untreated active hepatitis B
* Subjects have active hepatitis B

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 Weeks
  Objective Response Rate at 6 months using RECIST1.1 criteria

SECONDARY OUTCOMES:
Duration Response Rate | 6 Weeks
  ime from the date of the first documented response (CR or PR) to the earliest date of disease progression (RECIST 1.1), or death due to any cause.
Progression-free Survival | 6 Weeks
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause)
Overall Survival | 6 Weeks
  Time from enrollment until death due to any cause
incidence, type and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (about 24 months)
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: CongHua Xie, MD, Principal Investigator — Wuhan University; You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No